CLINICAL TRIAL: NCT03263260
Title: Prospective, Multicentric, Post-marketing Registry of Inspiron Sirolimus Eluting Coronary Stent for Treatment of Patients With Native Coronary Artery Lesions (Inspiron Real Life II)
Brief Title: Post-marketing Registry of Inspiron Sirolimus Eluting Coronary Stent
Acronym: Inspiron RL II
Status: Completed | Type: Observational
Sponsor: Scitech Produtos Medicos Ltda (Industry)
Responsible Party: Sponsor
Other Study IDs: Inspiron RL II
Record Dates: First submitted 2017-08-24; First posted 2017-08-28 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Coronary Artery Disease
Keywords: stent, DES, Inspiron
MeSH Terms: conditions — Coronary Artery Disease; Dysequilibrium syndrome | interventions — Mutagenesis, Insertional

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- implanted patients: Patients with native coronary artery lesions with diameter between 2.5 and 4.0 and 34 mm of length treated only with the Inspiron Sirolimus eluting Stent
  Interventions: Device: implant

INTERVENTIONS:
Device: implant — coronary stent implantation

SUMMARY:
Post-marketing, prospective, multicentric, non-randomized registry to evaluate the safety and efficacy of Inspiron Sirolimus Eluting Coronary Stent at the treatment of "real-world" patients.

DETAILED DESCRIPTION:
Up to 5.0000 patients with native coronary arteries lesions with diameter between 2.5 and 4.0 mm and 34 mm of length treated solely with the Inspiron Sirolimus Eluting Coronary Stent.

Stent implantation should be performed according to the Instructions for Use and according to the local practice. It is recommended that ECG and cardiac enzymes are collected before and after procedure. Dual anti-platelet therapy is recommended for at least 6 months after procedure.

Patients will be followed at 30 days, 1 and 2 years after procedure.

ELIGIBILITY:
Inclusion Criteria:

* alll patients that have been treated with the Inspiron Sirolimus Eluting Stent older and 18 years

Exclusion Criteria:

* Safein Vein or Left Internal Mammary artery Grafts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years submitted to implant of the Inspiron Sirolimus Eluting Stent in native coronary arteries
Sampling Method: Non-Probability Sample
Enrollment: 2504 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2024-01-21 (Actual)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events Rate | 12 months
  Cardiac Death, MI, Target Lesion Revascularization and Stent Thrombosis

SECONDARY OUTCOMES:
Target Vessel and Lesion Revascularization Rates | 24 months
  Target Vessel and Lesion Revascularization
Stent Thrombosis Rate | 24 months
  Stent Thrombosis

CONTACTS AND LOCATIONS:
Locations (1):
- União Brasileira de Educação e Assistência - Hospital São Lucas da PUC - RS, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No